CLINICAL TRIAL: NCT05553366
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of VX-548 for Acute Pain After a Bunionectomy
Brief Title: Evaluation of Efficacy and Safety of VX-548 for Acute Pain After a Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX22-548-104
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo matched to suzetrigine (SUZ) and hydrocodone bitartrate/acetaminophen (HB/APAP) for 2 days.
  Interventions: Drug: Placebo (matched to SUZ); Drug: Placebo (matched to HB/APAP)
- Hydrocodone bitartrate/acetaminophen (HB/APAP) (Active Comparator): Participants received HB 5 milligrams (mg)/ APAP 325 mg every 6 hours (q6h) for 2 days.
  Interventions: Drug: HB/APAP; Drug: Placebo (matched to SUZ)
- Suzetrigine (SUZ) (Experimental): Participants received SUZ [100 mg as first dose, followed by 50 mg every 12 hours (q12h)] for 2 days.
  Interventions: Drug: SUZ; Drug: Placebo (matched to HB/APAP)

INTERVENTIONS:
Drug: SUZ — Tablets for oral administration.
  Other Names: VX-548
  Arms: Suzetrigine (SUZ)
Drug: HB/APAP — Capsules for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP)
Drug: Placebo (matched to SUZ) — Placebo matched to SUZ for oral administration.
  Arms: Hydrocodone bitartrate/acetaminophen (HB/APAP); Placebo
Drug: Placebo (matched to HB/APAP) — Placebo matched to HB/APAP for oral administration.
  Arms: Placebo; Suzetrigine (SUZ)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of suzetrigine for acute pain after a bunionectomy.

ELIGIBILITY:
Key Inclusion Criteria:

* Before Surgery

  * Participants scheduled to undergo a primary unilateral bunionectomy with distal first metatarsal osteotomy (i.e., Austin procedure) and internal fixation under regional anesthesia (Mayo and popliteal sciatic block)
* After Surgery

  * Participant is lucid and able to follow commands
  * All analgesic guidelines were followed during and after the bunionectomy

Key Exclusion Criteria:

* Before Surgery

  * Prior history of bunionectomy or or other foot surgery on the index foot; or bunionectomy on the opposite foot
  * History of cardiac dysrhythmias within the last 2 years requiring anti-arrhythmia treatment(s)
  * Any prior surgery within 1 month before the first study drug dose
* After Surgery

  * Participant had a type 3 deformity requiring a base wedge osteotomy, concomitant surgery such as hammertoe repair; or experienced medical complications during the bunionectomy
  * Participant had a medical complication during the bunionectomy that, in the opinion of the investigator, should preclude randomization

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Shoals Medical Trials Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Trovare Clinical Research, Bakersfield, California
  - Pacific Research Network Inc, San Diego, California
  - New Hope Research Development, Tarzana, California
  - New Hope Research Development, West Covina, California
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Kansas Spine and Specialty Hospital, Wichita, Kansas
  - Midwest Clinical Research Center, Dayton, Ohio
  - Center for Orthopaedic Reconstruction and Excellence, Jenks, Oklahoma
  - HD Research LLC | First Surgical Hospital, Bellaire, Texas
  - HD Research LLC | Legent Orthopedic Hospital, Carrollton, Texas
  - HD Research LLC | Houston Heights Hospital, Houston, Texas
  - Futuro Clinical Trials, McAllen, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Houston Physicians Hospital, Webster, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Started | 216 | 431 | 428
Safety Set (Safety Set included all participants who received at least 1 dose of the study drug.) | 216 | 431 | 426
Completed | 208 | 419 | 418
Not Completed | 8 | 12 | 10
Not completed — Withdrawal of Consent (not due to AE | 4 | 8 | 5
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Other non-compliance | 1 | 1 | 0
Not completed — Randomized but not dosed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received placebo matched to SUZ and HB/APAP for 2 days.
- Hydrocodone Bitartrate/Acetaminophen (HB/APAP): Participants received HB 5 mg/ APAP 325 mg q6h for 2 days.
- Suzetrigine (SUZ): Participants received SUZ [100 mg as first dose, followed by 50 mg q12h] for 2 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ) | Total
Number analyzed (Participants) | 216 | 431 | 426 | 1073
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (13.5) | 48.3 (12.6) | 47.7 (13.3) | 48.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 359 | 366 | 912
  Male | 29 | 72 | 60 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 149 | 131 | 364
  Not Hispanic or Latino | 132 | 282 | 295 | 709
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 160 | 314 | 285 | 759
  Black or African American | 48 | 96 | 116 | 260
  Asian | 8 | 7 | 9 | 24
  American Indian or Alaska Native | 0 | 7 | 4 | 11
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1 | 2
  Other | 0 | 2 | 3 | 5
  Multiracial | 0 | 3 | 6 | 9
  Missing | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) From 0 to 48 Hours (SPID48), SUZ Compared to Placebo
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated subtracting the baseline pain intensity score from the pain intensity score at each postdose time point (using pain rating score range: 0= no pain to 10= worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours After First Dose of Study Drug
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
units on a scale | 70.6 (6.3) | 99.9 (4.5)
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0002, ANCOVA

2. Secondary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) as Recorded on a Numeric Pain Rating Scale (NPRS) From 0 to 48 Hours (SPID48), SUZ Compared to HB/APAP
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the baseline pain intensity score from the pain intensity score at each post dose time point(using pain rating score range: 0= no pain to 10= worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours After First Dose of Study Drug
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 431 | 426
units on a scale | 120.1 (4.5) | 99.9 (4.5)
Statistical Analysis 1: Comparison: Hydrocodone Bitartrate/Acetaminophen (HB/APAP) vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0016, ANCOVA

3. Secondary Outcome: Time to Greater Than or Equal to (≥)2-Point Reduction in NPRS,SUZ Compared to Placebo
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The time to ≥ 2-point reduction in NPRS from baseline was the time elapsed from the first dose of study drug until the first time the participant had at least a 2-point reduction in NPRS scores from baseline.
Time Frame: From Baseline Up to 48 Hours After First Dose of Study Drug
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure. Data for this outcome measure was planned to be collected and analyzed only for the Placebo and SUZ group.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
minutes | 480 [476 to 716] | 240 [117 to 477]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0016, Log Rank

4. Secondary Outcome: Time to ≥1-Point Reduction in NPRS, SUZ Compared to Placebo
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The time to ≥1-point reduction in NPRS from baseline was the time elapsed from the first dose of study drug until the first time the participant had at least a 1-point reduction in NPRS from baseline.
Time Frame: From Baseline Up to 48 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
minutes | 61 [34 to 121] | 60 [58 to 65]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.1315, Log Rank

5. Secondary Outcome: Percentage of Participants Reporting Good or Excellent on the Patient Global Assessment (PGA) Scale, SUZ Compared to Placebo
Description: The PGA is a single-item assessment of patient perceptions of the method of pain control with the study drug and is evaluated on a 4-point Likert scale as: (poor, fair, good, or excellent). Percentage of participants who reported good or excellent on the PGA scale were reported.
Time Frame: At 48 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
percentage of participants | 53.2 | 61.7
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0343, Cochran-Mantel-Haenszel

6. Secondary Outcome: Incidence of Vomiting or Nausea, SUZ Compared to HB/APAP
Description: The percentage of participants with the events of vomiting or nausea during the specified time frame was reported.
Time Frame: From Baseline up to Day 19
Population: Safety Set included all participants who received at least 1 dose of study drug. Data for this outcome measure was planned to be collected and analyzed only for the HB/APAP and SUZ group.
Measure: Number; unit: percentage of participants
Arm/Group | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 431 | 426
percentage of participants | 16.5 | 9.2
Statistical Analysis 1: Comparison: Hydrocodone Bitartrate/Acetaminophen (HB/APAP) vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0014, Pearson's chi-squared test

7. Secondary Outcome: Time-weighted SPID as Recorded on the NPRS From 0 to 24 Hours (SPID24), SUZ Compared to Placebo
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the baseline pain intensity score from the pain intensity score at each post dose time point (using pain rating score range: 0= no pain to 10= worst possible pain). SPID24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
units on a scale | 19.8 (3.0) | 30.6 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0032, ANCOVA

8. Secondary Outcome: Time to First Use of Rescue Medication, SUZ Compared to Placebo
Description: Time to first use of rescue medication is the time from the first dose of study drug until the first use of rescue medication.
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
minutes | 185 [143 to 210] | 157 [145 to 192]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.8592, Log Rank

9. Secondary Outcome: Percentage of Participants Using Rescue Medication From 0 to 48 Hours, SUZ Compared to Placebo
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
percentage of participants | 85.6 | 85.4
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.9143, Cochran-Mantel-Haenszel

10. Secondary Outcome: Total Rescue Medication Usage, SUZ Compared to Placebo
Time Frame: 0 to 48 Hours After First Dose of Study Drug
Population: as for outcome 3
Measure: Median (Full Range); unit: milligram
Arm/Group | Placebo | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 426
milligram | 800 [0 to 3200] | 800 [0 to 3200]
Statistical Analysis 1: Comparison: Placebo vs Suzetrigine (SUZ); Test type: Superiority; p = 0.0205, Wilcoxon rank-sum

11. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Day 19
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
Number analyzed (Participants) | 216 | 431 | 426
Participants
  Participants with TEAEs | 76 | 180 | 132
  Participants with SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 19
Description: Safety Set included all participants who received at least 1 dose of the study drug.
Arm/Group | Placebo | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Suzetrigine (SUZ)
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/431 | 0/426
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/431 | 0/426
Other Adverse Events (participants affected / at risk) | 51/216 | 113/431 | 72/426
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=216) | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) (N=431) | Suzetrigine (SUZ) (N=426)
Constipation (Gastrointestinal disorders) | 9 | 22 | 15
Nausea (Gastrointestinal disorders) | 23 | 62 | 35
Dizziness (Nervous system disorders) | 11 | 23 | 15
Headache (Nervous system disorders) | 20 | 45 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05553366/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT05553366/SAP_001.pdf